CLINICAL TRIAL: NCT01529944
Title: Genetic Testing of Noonan Subjects Previously Treated With Norditropin® in the GHNOO-1658 Trial
Brief Title: Genetic Testing of Noonan Subjects Previously Treated With Norditropin®. An Extension to Trial GHNOO-1658
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHNOO-3680; 2008-004535-38 (EudraCT Number)
Record Dates: First submitted 2012-01-02; First posted 2012-02-09 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Genetic Disorder; Noonan Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Noonan Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose 33 mcg/kg/day (Experimental)
  Interventions: Drug: somatropin
- High dose 66 mcg/kg/day (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Results from a genetic testing for the PTPN11 mutation will be collected retrospectively for 24 subjects with Noonan syndrome previously treated with somatropin in accordance with the S/GHD/004/N00 protocol and in the follow-up trial GHNOO-1658.
  Arms: Low dose 33 mcg/kg/day
Drug: somatropin — Results from a genetic testing for the PTPN11 mutation will be collected retrospectively for 24 subjects with Noonan syndrome previously treated with somatropin in accordance with the S/GHD/004/N00 protocol and in the follow-up trial GHNOO-1658.
  Arms: High dose 66 mcg/kg/day

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to obtain the PTPN11 mutation status and investigate the impact of the PTPN11 mutation status on the effect of somatropin (Norditropin®) by use of data obtained in the GHNOO-1658 trial.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the GHNOO-1658 trial
* Subject has completed genetic testing of PTPN11 mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Change in height SDS (Standard Deviation Score) (referenced to normal population) | From baseline until final height is reached

SECONDARY OUTCOMES:
Final height SDS (referenced to normal population) | From baseline until final height is reached
Final height SDS (referenced to Noonan population) | From baseline until final height is reached
Change in height SDS (referenced to Noonan population) | From baseline until final height is reached
Number of subjects with final height SDS above - 2SDS (reference to normal population) | When final height is reached
Proportion of subjects with final height SDS above - 2SDS (reference to normal population) | When final height is reached
Adverse events | From baseline until final height is reached

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Gothenburg, Sweden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com